CLINICAL TRIAL: NCT07367958
Title: A Phase 1, Randomized, Open-label, Two-arm, Parallel-Group, Single-dose Study to Compare Pharmacokinetics and Safety of CT-P52 AI and CT-P52 PFS in Healthy Male Subjects
Brief Title: A Study to Compare the Auto-injector and Pre-filled Syringe of CT-P52 in Healthy Male Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CT-P52 1.2
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P52 Auto-injector (Experimental): CT-P52, 80 mg in 1 ml, a single subcutaneous (SC) injection via auto-injector (AI)
  Interventions: Biological: CT-P52
- CT-P52 Pre-filled syringe (Active Comparator): CT-P52, 80 mg in 1 ml, a single SC injection via pre-filled syringe (PFS)
  Interventions: Biological: CT-P52

INTERVENTIONS:
Biological: CT-P52 — CT-P52, 80 mg in 1 ml, a single subcutaneous (SC) injection via auto-injector (AI)

SUMMARY:
This is phase 1 study to Compare the Pharmacokinetics, Safety and Immunogenicity of the Auto-injector and Pre-filled syringe of CT-P52 in Healthy Male Subjects.

DETAILED DESCRIPTION:
CT-P52, containing the active ingredient ixekizumab, is being developed by CELLTRION, Inc. as a proposed biosimilar to the reference product, Taltz. In this study, Pharmacokinetics, Safety and Immunogenicity of the Auto-injector and Pre-filled syringe of CT-P52 will be evaluated in Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, between the ages of 19 and 55 years, both inclusive.
* Subject has a body weight between 60 to 90 kg, both inclusive, and a BMI between 18.0 and 29.9 kg/m2, both inclusive, when rounded to the nearest tenth.

Exclusion Criteria:

* A medical history and/or condition that is considered significant
* Clinically significant allergic reactions, hypersensitivity
* History or current infection of hepatitis B virus, hepatitis C virus, human immunodeficiency virus, or syphilis
* Active or latent Tuberculosis
* History of malignancy
* Previous exposure to ixekizumab or a biosimilar of ixekizumab or any drug that directly targets Interleukin (IL)-17 or the IL-17 receptor

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
PK similarity demonstration by AUC 0-inf | Day 85
  Demonstrate the PK similarity in terms of area under the concentration-time curve from time zero to infinity (AUC0-inf) of CT-P52 SC administration via AI versus PFS in healthy male subjects up to Day 85.
PK similarity demonstration by Cmax | Day 85
  Demonstrate the PK similarity in terms of maximum serum concentration (Cmax) of CT-P52 SC administration via AI versus PFS in healthy male subjects up to Day 85.

SECONDARY OUTCOMES:
Additional PK evaluation by AUC0-last | Day 85
  Evaluate additional PK in terms of AUC from time zero to the last quantifiable concentration (AUC0-last).
Additional PK evaluation by Tmax | Day 85
  Evaluate additional PK in terms of time to maximum concentration (Tmax).
Additional PK evaluation by T1/2 | Day 85
  Evaluate additional PK in terms of terminal half-life (t1/2).
Additional PK evaluation by %AUCext | Day 85
  Evaluate additional PK in terms of percentage of area under the concentration-time curve from time zero to infinity (AUC0-inf) obtained by extrapolation (%AUCext).
Safety evaluation by AEs | Day 85
  Evaluate safety in terms of adverse events (including treatment-emergent adverse events [TEAEs] and serious adverse events[SAEs]).

IPD SHARING:
Plan to Share IPD: No